CLINICAL TRIAL: NCT06338306
Title: Therapeutic Drug Monitoring of Tacrolimus Personalized Therapy in Heart Transplantation: New Strategies
Brief Title: Tacrolimus and Personalized Therapy to Prevent Acute Rejection Episodes
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: 08073421
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Heart Transplant Failure
Keywords: Tacrolimus; Whole Blood; PBMCs; Endomyocardial biopsy; Acute rejection; Therapeutic Drug Monitoring (TDM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- De novo heart transplant patients: Twenty-five de-novo heart transplant recipients will be enrolled, male and female, aging 18-70 years, receiving TAC in combination with steroids and antiproliferative drugs (MMF; EC-MPS) or m-TOR inhibitors (Everolimus; Sirolimus).
  Interventions: Drug: Tacrolimus（FK506）

INTERVENTIONS:
Drug: Tacrolimus（FK506） — Prograf

SUMMARY:
Heart transplant is the only effective treatment for people with advanced heart failure.

Post-transplant pharmacological therapies are of fundamental importance for the survival of individuals after surgery: although considerable progress has been made for combined immunosuppressive therapies, acute cellular and especially non-cellular rejection still represents a great challenge for doctors.

To verify the absence of the first signs of acute rejection, the analysis of numerous cardiac biopsies (EMB endomyocardial biopsies) is necessary during the first 12 months following the transplant.

Thanks to these scheduled checks, doctors are able to identify the first symptoms of possible chronic rejection and reduce its episodes.

Since the analysis of biopsies is also based on subjective interpretations, cases of erroneous conclusions are frequent.

The researchers of this study aim not only to analyze the biopsies according to the current best clinical practice, but also to evaluate how much anti-rejection drug is actually contained within them.

This is an analysis that is still little used for this type of transplant, which could provide very useful information to doctors.

The researchers will focus their attention on one drug in particular, tacrolimus, abbreviated to "TAC".

The amount of drug measured in biopsies will be compared with that measured in whole blood samples and in particular blood cells (peripheral blood mononuclear cells: PBMC).

The genetic characteristics of each person play an important role in the success of treatment with the drug. To best interpret the results, all participants will be asked to take a blood sample to identify some characteristics of their DNA that could influence the outcome of tacrolimus therapy.

DETAILED DESCRIPTION:
Heart transplant is the only effective treatment for people with advanced heart failure. Major advances in allograft protection, such as improved combined immunosuppressive therapies, have led to progressive increases in post-transplant survival, but acute cellular and especially non-cellular rejection still represents a challenge for clinicians. Endomyocardial biopsy (EMB) is the current standard of care used to identify rejection after HTx, with at least 13 biopsies scheduled within the twelve months following transplantation.

The mortality rate, after this period, is approximately 3.5% per year and the causes of death range from primary graft failure and multiorgan failure, to neoplasms, renal failure and cardiac allograft vasculopathy. Although acute rejection can be well managed in most cases, episodes of cumulative rejection and chronic rejection are likely to contribute to long-term graft failure and graft vasculopathy. The current ISHLT (International Society for Heart and Lung Transplantation) classification system provides categories of severity of rejection, for both cellular and antibody-mediated rejection. It describes the degree of tissue damage and infiltration by inflammatory cells and states that the greater the infiltrate, the worse the rejection. The purpose of the evaluation is to guide doctors in treating rejection before symptoms appear. However, histological reading, like any diagnostic technique, is subject to false positives and false negatives.

The researchers propose to monitor TAC trough concentrations directly in EMBs, during the first year after transplantation (5 scheduled biopsies), from at least 25 de novo heart transplant recipients. The results will be analyzed and correlated with whole blood and with the minimum concentrations of PBMC (peripheral blood mononuclear cells) detected, for each patient, in the same 5 scheduled follow-up visits. Pharmacogenetic studies will focus on CYP3A4, CYP3A5 and ABCB1 gene variants. The ABCB1 gene encodes P-glycoprotein (Pg-p), an ATP-driven transmembrane transporter that acts as an efflux pump and transports TAC out of PBMCs and tissues. These researchers hypothesize that elevated cardiac expression of P-gp may reduce TAC uptake into cardiac (donor) tissue, may act as an important modulator of immunosuppressive effects, and thus have important therapeutic implications.

Main objectives

Tacrolimus is a critically dosed drug and therapeutic drug monitoring is mandatory to avoid under- and overexposure. However, rejection and drug-related toxicity occur despite pre-dose whole blood (blood [TAC]) tacrolimus concentrations being on target. Monitoring tacrolimus concentrations at the target site (within peripheral blood mononuclear cells ([TAC] cells)) and directly in endomyocardial biopsies ([TAC] EMB)) may better correlate with treatment efficacy.

The objectives of this study are:

1. study TAC trough concentrations in whole blood (blood [TAC]), PBMC (cells [TAC]), and EMB ([TAC]EMB) simultaneously, across 5 scheduled follow-up visits of 25 HTx recipients
2. identify genetic characteristics that influence the metabolism and distribution of tacrolimus in whole blood, cells and EMBs,
3. study the relationships between the three concentration profiles ([TAC]blood), [TAC]cells, [TAC]EMB) and clinical outcomes, during the first year after heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

de novo heart transplant recipient

Exclusion Criteria:

* Age < 18 years
* Intolerance to TAC or to some excipient
* Intolerance to glucose
* diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Twenty-five de-novo heart transplant recipients will be enrolled, male and female, aging 18-70 years, receiving TAC in combination with steroids and antiproliferative drugs (MMF; EC-MPS) or m-TOR inhibitors (Everolimus; Sirolimus).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tacrolimus quantification in an unconventional matrix | 0.5, 1, 3, 6 and 12 months after heart transplantation
  Each biopsy will be weighed immediately after being taken from the transplanted organ during the 5 scheduled follow up visits.
  Tacrolimus will be extraxcted following a validated and published alalytical procedure, consisting of a combined enzymatic-digestion/mass spectrometry assay (online SPE-LC-MS/MS).
  Enzymatic tissue digestion followed by a liquid-liquid drug extraction in the same vial of reaction will allow us to avoid both sample loss and contaminations.
  TAC concentrations will be expressed as "pg TAC/mg biopsy"
Tacrolimus quantification in PBMCs | 0.5, 1, 3, 6 and 12 months after heart transplantation
  10 mL of peripheral blood will be collected and processed by Fycoll gradient procedure for the PBMCs separation.
  PBMCs will be isolated and then counted with an automated cell counter.
  TAC concentration in PBMCs (expressed as "ng/1.000.000 cells") will be detected by a validated online SPE- LC-MS/MS method.
Tacrolimus quantification in whole blood | 0.5, 1, 3, 6 and 12 months after heart transplantation
  The TAC concentration will be detected in whole blood using an automatic immunoassay system, used daily for routine monitoring.
  TAC concentration will be expressed as "ng/mL" in whole blood.
  Therapeutic range: 5-20 ng/mL

SECONDARY OUTCOMES:
Genetic profile in heart transplant recipients | The pharmacogenetic investigation (PGx) will be carried out at enrollment
  Variants in the CYP3A4, CYP3A5 and ABC1 will be analyzed:
  CYP3A4*22 (SNP rs35599367: 522-191C> T) CYP3A5*3 (rs776746, 6986A> G) CYP3A5*1 The most frequently studied polymorphisms in the ABCB1 gene are C1236T (rs1128503), G2677T/A (rs2032582) and C3435T (rs1045642).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molinaro M, Pellegrini C, Cattadori B, De Gregori S. Development and validation of a combined enzymatic-digestion/mass spectrometry assay for Tacrolimus quantitation in cardiac biopsies. J Chromatogr B Analyt Technol Biomed Life Sci. 2020 Sep 1;1152:122215. doi: 10.1016/j.jchromb.2020.122215. Epub 2020 Jun 21. PMID 32615534